CLINICAL TRIAL: NCT05729971
Title: Nasogastric Tube After Laparoscopic Heller-Dor Myotomy: do You Really Need it?
Brief Title: Nasogastric Tube After Laparoscopic Heller-Dor Myotomy
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Giuseppe Palomba, M.D, PhD student, Federico II University
Other Study IDs: 292/190
Record Dates: First submitted 2023-01-27; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Achalasia; Achalasia Cardia
Keywords: Heller Laparoscopic; Dor Laparoscopic
MeSH Terms: conditions — Esophageal Achalasia | interventions — Enteral Nutrition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- with NGT: In these patients, the nasogastric tube remains after surgery. It was removed after x-ray test.
  Interventions: Procedure: nasogastric tube
- noNGT: In these patients, NGT was removed at the end of surgery.

INTERVENTIONS:
Procedure: nasogastric tube — The intervention consists in removing or not the nasogastric tube at the end of the surgery.
  Groups: with NGT

SUMMARY:
The goal of this prospective observational study is to evaluate the role of nasogastric tube (NGT) in patients with achalasia underwent to Heller-Dor laparoscopic. The main question it aims to answer are:

• If it is possible to remove NGT at the end of surgery. Participants will be dived in two groups: the first one with NGT after surgery and second one without NGT (noNGT).

If there is a comparison group: Researchers will compare group NGT and group noNGT to see if routine placement of NGT is useless.

DETAILED DESCRIPTION:
Achalasia is a rare disease characterized by dysfunction of low oesophageal sphincter. This disease is divided according to Chicago classification into three subtypes.

Laparoscopic Heller - Dor is a important treatment of types I and II Achalasia. There are several studies evaluating the NGT in colorectal, hepatic, urologic, thoracic, otorhinolaryngology, gastric and esophageal surgery. Its use in postoperative period in achalasic patients is not yet clear.

Historically, NGT has been used to reduce gastric distention, nausea, vomiting and chest pain.

The aim of our study is to value the role of NGT for this surgery. We prospectively enrolled achalasic patients undergoing laparoscopic Heller -Dor .

The NGT group and noNGT were compared in terms of perioperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* patients with achalasia of type I and II
* patients undergoing laparoscopic Heller-Dor
* patients older than 18 years
* both sexes

Exclusion Criteria:

* pregnant patients;
* patients a history of abdominal surgery;
* body mass index (BMI) >40;
* American Society of Anesthesiology (ASA) score >4;
* megaesophagus;
* III type Achalasia;
* previously treated for this disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Each patient has type I or type II esophageal achalasia and was treated with the Heller-Dor laparoscopic surgery.
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Nausea | in the first postoperative day
  clinically evaluating the presence or absence
vomiting | in the first postoperative day
  clinically evaluating the presence or absence
chest pain | in the first postoperative day
  clinically evaluating the presence or absence

SECONDARY OUTCOMES:
Length of stay | from the first postoperative day to the third postoperative day
  days of hospitalization from first postoperative day
First flatus | from the first postoperative day to the third postoperative day
  on which postoperative day the patient had the first flatus.
Intake liquid diet | from the first postoperative day to the third postoperative day
  when the patient starts drinking
Intake semi-solid diet (day) | from the first postoperative day to the third postoperative day
  when the patient starts to eat
postoperative complications | from the first postoperative day to the third postoperative day
  Based on Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Aprea, professor, Study Director — Federico II University
Locations (1):
- AOU. policlinico, Federico II, Napoli, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Patients Number Length of stay (day) First flatus (day) Intake liquid diet (day) Intake semi-solid diet (day) Intraoperative complications
  Postoperative complications:
  * Grade I
  * Grade II

REFERENCES:
- [Background] Hoshino M, Omura N, Yano F, Tsuboi K, Kashiwagi H, Yanaga K. Immunohistochemical study of the muscularis externa of the esophagus in achalasia patients. Dis Esophagus. 2013 Jan;26(1):14-21. doi: 10.1111/j.1442-2050.2011.01318.x. Epub 2012 Feb 6. PMID 22309323
- [Background] Andolfi C, Fisichella PM. Meta-analysis of clinical outcome after treatment for achalasia based on manometric subtypes. Br J Surg. 2019 Mar;106(4):332-341. doi: 10.1002/bjs.11049. Epub 2019 Jan 28. PMID 30690706
- [Background] Arcerito M, Jamal MM, Perez MG, Kaur H, Sundahl A, Moon JT. Esophageal Achalasia: From Laparoscopic to Robotic Heller Myotomy and Dor Fundoplication. JSLS. 2022 Jul-Sep;26(3):e2022.00027. doi: 10.4293/JSLS.2022.00027. PMID 35967962